CLINICAL TRIAL: NCT06289699
Title: Alert Frequency, Nurse, and Patient Satisfaction With a Continuous Wireless Vital Sign Monitoring Software Across Health Care Systems and Cultures
Brief Title: Alert Frequency, Nurse, and Patient Satisfaction With a wCVSM Software Across Health Care Systems and Cultures
Status: Recruiting | Type: Observational
Sponsor: Christian S. Meyhoff (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Christian S. Meyhoff, Professor, PhD, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Other Study IDs: WARD-CSS international 1251
Record Dates: First submitted 2024-01-22; First posted 2024-03-04 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: User Experience; Postoperative Complications; Acute Medical Conditions
Keywords: continuous wireless vital sign monitoring; vital sign deviation; healthcare system and culture; User Experience; Postoperative Complications; Acute Medical Conditions
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this prospective, international multi-centre pilot study is to assess the functionality and user experience of a new vital sign monitoring system in 20 patients and 20 nurses in the general ward at each centre. The patients will be monitored with a wireless, continuous vital sign monitoring systems and answer a questionnaire afterwards. They will in addition have vital signs monitored as per standard practice. The nurses will answer a questionnaire after having had the responsibility for a monitored patient for a full shift. The main aims are: To determine the frequency of alerts activated in the app in relation to the alerts that should be activated based on measured data, to explore current practices of in-hospital monitoring by semi-structured interviews to map differences across systems and to test nurse and patient satisfaction.

DETAILED DESCRIPTION:
The participants will be monitored for 4 days postoperatively or for 4 days after acute admission and until discharge.

Monitoring devices used in this study will be validated FDA or/and CE approved devices used within their original purpose. Centers can choose to use Sotera Visimobile or Isansys Lifeguard with accompanying sensors. These devices will be used together with the CE approved WARD web and mobile application.

Study sites include: St. Olav Hospital Trondheim, Royal Liverpool University Hospital, University Medical Centre Hamburg-Eppendorf,University Medical Centre Groningen, The Netherlands and the Cleveland Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Expected stay in the hospital ≥2 days
* Admitted for surgery with expected duration of surgery >2 hours or admitted for acute medical condition with at least one of the following vital sign deviations within 24 hours of acute admission, recorded by the staff

  * RR > 21 breaths pr minute
  * RR < 11 breaths pr minute
  * Pulse (P) > 91 beats pr minute
  * Pulse (P) < 50 beats pr minute
  * SpO2 < 94 % without oxygen supplementation
  * Systolic BP < 110 mmHg
  * Systolic BP > 220 mmHg

Exclusion Criteria:

* Participant expected not to cooperate with study procedures.
* Allergy to plaster or silicone.
* Pacemaker or Implantable Cardioverter Defibrillator (ICD) device.
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 Patients in the general ward (surgical or medical) will be monitored with wCVSM and answer a questionnaire afterwards. 20 nurses will answer a questionnaire after having had the responsibility for a monitored patient for a full shift (including a shift where monitoring is initiated or a shift where the patient is discharged). Therefore, multiple nurses can be interviewed per patient. Patients will in addition have vital signs monitored as per standard practice. Participants will be recruited from wards at the study sites.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of alerts activated in the app in relation to the alerts that should be activated based on measured data | during monitoring period, on average 3 months

SECONDARY OUTCOMES:
Technical feasibility | during monitoring period, on average 3 months
  will be assessed as data capture of vital signs as percentage of data from each of the vital sign sensors of the total monitoring period.
Alert relay to smartphones | during monitoring period, on average 3 months
  will be assessed by comparing % of alerts received compared to alerts generated by the WARD24/7 App.
Response to alerts | during monitoring period, on average 3 months
  will be assessed using the response buttons as % of nurses pressing attend, snooze, or refer to colleague on the WARD24/7 App.
Patients experiences from being monitored with wCSVM. | during monitoring period, on average 3 months
  will be assessed by a questionnaire named "Patient experience with wireless vital sign monitorering" consisting of 8 items. Each item can be answered with: strongly agree, agree, neither agree nor disagree, disagree, and strongly disagree.
Relevance of alarms | during monitoring period, on average 3 months
  by using feedback from the nurses given in the app, % of relevant alerts
Frequency of delivered alarms on oxygen saturation (SpO2) pr patient pr day | during monitoring period, on average 3 months
Frequency of delivered alarms on respiration rate (RR) pr patient pr day | during monitoring period, on average 3 months
Frequency of delivered alarms on heart rate (HR) pr patient pr day | during monitoring period, on average 3 months
Frequency of delivered alarms on blod pressure (BP) pr patient pr day | during monitoring period, on average 3 months
Overall score of user satisfaction from use of WARD24/7 app | during monitoring period, on average 3 months
  assessed by the mHealth App Usability Questionnaire (MAUQ) consisting of 18 items. In this questionnaire, 1 - strongly disagree, 2 - disagree, 3 - somewhat disagree, 4 - neither agree nor disagree, 5 - somewhat agree, 6 - agree, 7 - strongly agree.To determine the usability of an app, calculate the total and determine the average of the responses to all statements. The higher the overall average, the higher the usability of the app.
Subscale MAUQ scores | during monitoring period, on average 3 months
  assessed by the mHealth App Usability Questionnaire (MAUQ) consisting of 18 items. In this questionnaire, 1 - strongly disagree, 2 - disagree, 3 - somewhat disagree, 4 - neither agree nor disagree, 5 - somewhat agree, 6 - agree, 7 - strongly agree.To determine the usability of an app, calculate the total and determine the average of the responses to all statements. The higher the overall average, the higher the usability of the app.
  Ease of use and satisfaction (5 items, MAUQ_E), system information arrangement (7 items, MAUQ_I), and usefulness (6 items, MAUQ_U).
Monitoring practices prior to the wCVSM | Baseline, on average 3 months
  assessed by a semi structured interview guide including information on type of monitoring (manual/intermittent, type of vital signs collected, frequency of measurements, escalation protocols etc.).

OTHER OUTCOMES:
Cumulative duration of SpO2<88% and SpO2 < 85% | during monitoring period, on average 3 months
Cumulative duration of respiratory rate ≤ 5 min-1 and Respiratory rate > 24 min-1 | during monitoring period, on average 3 months
Cumulative duration of Heart rate > 130 min-1 and Heart rate ≤ 30 min-1 | during monitoring period, on average 3 months
Cumulative duration of Systolic blood pressure ≤ 90 mmHg and Systolic blood pressure > 220 mmHg o | during monitoring period, on average 3 months
Cumulative duration of Circulatory failure | during monitoring period, on average 3 months
Cumulative duration of Systolic blood pressure ≤ 90 mmHg AND Heart rate >110 min-1 OR heart rate < 50 bpm AND/OR SpO2 < 92% o | during monitoring period, on average 3 months
Cumulative duration of Hypoventilation: RR < 11 AND SpO2 < 88% | during monitoring period, on average 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Meyhoff, MD, PhD, Principal Investigator — Copenhagen University Hospital - Bispebjerg and Frederiksberg, Copenhagen, Denmark; Eske K Aasvang, MD, DMSci, Principal Investigator — Rigshospitalet, Copenhagen University, Copenhagen, Denmark
Locations (5):
- The Cleveland Clinic Foundation, General Anesthesiology, Cleveland, Ohio, United States
- Universitätsklinikum Hamburg-Eppendorf (UKE), Zentrum für Anästhesiologie und Intensivmedizin, Klinik und Poliklinik für Anästhesiologie, Hamburg, Germany
- University Medical Center Groningen, Department of Anesthesiology, Groningen, Netherlands
- St. Olavs Hospital HF, Klinikk for anestesi og intensivmedisin, Trondheim, Norway
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No